CLINICAL TRIAL: NCT00555789
Title: A 24 Month Extension to a 12-month Open Label, Randomized, Multicenter Study Evaluating Efficacy, Safety and Tolerability of Oral AEB071 Plus Tacrolimus (Converted to Mycophenolic Acid After 3 Months), vs. Mycophenolic Acid Plus Tacrolimus in de Novo Renal Transplant Recipients
Brief Title: 24 Month Extension to Efficacy and Safety of AEB071 Plus Tacrolimus (Converted to Mycophenolic Acid After 3 Months) in Renal Transplant Patients(Converted to Mycophenolic Acid After 3 Months) in Renal Transplant Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEB071A2203E1
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-07

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; rejection; AEB071; tacrolimus; mycophenolic acid; immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — sotrastaurin; Tacrolimus

ARMS (2):
- 1 (Active Comparator): mycophenolic and tacrolimus
  Interventions: Drug: mycophenolic plus tacrolimus
- 2 (Experimental): mycophenolic and tacrolimus
  Interventions: Drug: AEB071

INTERVENTIONS:
Drug: AEB071 — 200mg oral b.i.d.
  Other Names: mycophenolic plus tacrolimus
  Arms: 2
Drug: mycophenolic plus tacrolimus — 720mg b.i.d. 2yrs
  Arms: 1

SUMMARY:
This study will provide continued treatment and assess the long term safety, efficacy and tolerability of oral AEB071 plus tacrolimus vs. mycophenolic acid plus tacrolimus after kidney transplantation.

ELIGIBILITY:
Inclusion criteria:

* Participation in core study CAEB071A2203
* The patient has been maintained on AEB071/mycophenolic acid or tacrolimus/mycophenolic acid, consistent with their original randomization, at their core study Month 12 visit.
* Women capable of becoming pregnant are required to practice a medically approved method of birth control as long as they are on study medication and for a period of 3 months following discontinuation of study drug(s).

Exclusion criteria:

* Pregnancy. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Long term safety assessed by and renal safety defined by measuring renal function using Modification of Diet in Renal Disease (MDRD) formula for Glomerular Filtration Rate (GFR) beyond 12 months. | three Yrs

SECONDARY OUTCOMES:
Efficacy assessed by: the incidence over 36 months of the composite endpoint of biopsy proven rejection ≥ 1A, graft loss, death, or loss to follow-up in the two study arms. | Three yrs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (26):
- United States (2):
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Madison, Wisconsin
- Novartis Investigative Site, Halifax, Canada
- France (4):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
- Italy (3):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Padua
- Spain (4):
  - Novartis Investigative Site, Llobregat
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- United Kingdom (4):
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

REFERENCES:
- See also: Results for CAEB071A2203E1 on the Novartis clinical trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2800